CLINICAL TRIAL: NCT00903071
Title: Personalized Physician Learning Intervention to Improve Hypertension Care
Brief Title: Personalized Physician Learning to Improve Hypertension Care
Acronym: PPL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Collaborators: University of Minnesota (Other); Kaiser Permanente (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 07-090; R01HL089451-01A1 (NIH)
Record Dates: First submitted 2009-05-13; First posted 2009-05-15 (Estimated); Last update posted 2014-06-16 (Estimated); Status verified 2014-06

CONDITIONS: Hypertension
Keywords: Hypertension; Primary Care; Physician Learning
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- REAL PPL (Active Comparator): REAL+PPL profiles PCP performance using real electronic medical record derived data to identify each PCP's specific failures of decision making in HT care antecedent to the personalized learning intervention.
  Interventions: Behavioral: Real PPL
- SIM PPL (Active Comparator): SIM+PPL, profiles PCP performance using simulated cases to identify each PCP's specific failures of decision making in HT care antecedent to the personalized learning intervention.
  Interventions: Behavioral: Sim PPL
- Control (No Intervention): No intervention -control group

INTERVENTIONS:
Behavioral: Real PPL — See above arm description
  Arms: REAL PPL
Behavioral: Sim PPL — See above arm description
  Arms: SIM PPL

SUMMARY:
In this project the investigators implement and test the ability of a Personalized Physician Learning (PPL) intervention to improve hypertension (HT) care with the following specific aims:

Specific Aim 1: Implement two versions of a Personalized Physician Learning (PPL) intervention and assess the ability of these interventions to improve hypertension control in primary care practice.

* Hypothesis 1: Patients of physicians who receive the REAL+PPL Intervention (Group 1) will subsequently have better HT control compared to patients of control group physicians (Group 3).
* Hypothesis 2: Patients of physicians who receive the SIM+PPL Intervention (Group 2) will subsequently have better HT control compared to patients of control group physicians (Group 3).
* Hypothesis 3: Patients of physicians who receive the REAL+PPL (Group 1) will subsequently have better HT control compared to patients of physicians who receive the SIM+PPL (Group 2).

Specific Aim 2: Assess the cost-effectiveness of the SIM+PPL and REAL+PPL interventions, relative to no intervention.

DETAILED DESCRIPTION:
The objective of this project is to improve hypertension (HT) control by implementing two Personalized Physician Learning interventions designed for primary care physicians (PCPs). Improved HT control has long been identified as a major national health care priority because uncontrolled HT is a leading cause of stroke(CVA), congestive heart failure (CHF), chronic kidney disease (CKD), end-stage renal disease (ESRD),myocardial infarction (MI), and other adverse health events. The cost of uncontrolled HT and its sequelae is estimated to be at least $100 billion dollars a year in the U.S., and there has been only minimal improvement in HT care in recent decades. Currently, of an estimated 68 million Americans with HT, about 42 million remain uncontrolled.

Personalized Physician Learning (PPL) interventions are powerful enough to change physician behavior and improve HT care. The PPL interventions in this project are directed to individual primary care physicians(PCPs) using a simple 3-step approach: (a) Analyze each physician's pre-intervention patterns of HT care to identify specific failures of physician decision making in HT care, (b) Provide each physician with a series of personalized HT learning cases designed to correct the failures of decision making that result in that physician's observed patterns of HT care. Learning cases provide iterative on-screen feedback of blood pressure (BP) changes in response to a sequence of changes in therapy, expert-generated suggestions for better HT care, and adaptive selection of subsequent cases until identified errors in decision making are mastered. (c) Assess intervention impact on the care of actual patients with HT in the post-intervention period, to assess transfer of learning from the simulated to the office practice environment. The PPL intervention strategy is based on recent work in cognitive science and learning theory and has been successfully applied in other research and educational settings, although it has yet to be applied to HT care.

ELIGIBILITY:
Inclusion Criteria:

* Practicing physician at 1 of 2 medical groups.
* Be a general internist of family physician.
* Provide ongoing clinical care to at least 25 adult patients with uncontrolled hypertension. Additional patient criteria include;
* 22 years or more on date of physician randomization.
* Charlson score less than 4.
* Be linked to a primary care physician who has consented to the study.
* Have 2 consecutive office blood pressure readings above the 7th Report of the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure (JNC7) goal, within a 12 month time period.

Exclusion Criteria:

* Physicians practicing at a second clinic for more than 1 day per week. Additional patient criteria;
* Less than 22 years of age.
* Charlson score of >= 4

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2010-03; Primary Completion 2011-12 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Hypertension control | 12 month pre and 12 month post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Patrick J O'Connor, MD, MPH, Principal Investigator — HealthPartners Institute
Locations (1):
- HealthPartners Research Foundation, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] O'Connor PJ, Magid DJ, Sperl-Hillen JM, Price DW, Asche SE, Rush WA, Ekstrom HL, Brand DW, Tavel HM, Godlevsky OV, Johnson PE, Margolis KL. Personalised physician learning intervention to improve hypertension and lipid control: randomised trial comparing two methods of physician profiling. BMJ Qual Saf. 2014 Dec;23(12):1014-22. doi: 10.1136/bmjqs-2014-002807. Epub 2014 Sep 16. PMID 25228778